CLINICAL TRIAL: NCT02407717
Title: Venous Thromboembolism and Bleeding in Hospitalized Medical Patients With Cancer
Status: Completed | Type: Observational
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Marcello Di Nisio, Principal Investigator, G. d'Annunzio University
Other Study IDs: ChietiOnco2
Record Dates: First submitted 2015-03-20; First posted 2015-04-03 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Hemorrhage; Vein Thrombosis
MeSH Terms: conditions — Hemorrhage; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with cancer hospitalized for an acute medical illness have an increased risk of venous thromboembolic events. Although international guidelines suggest the use of thromboprophylaxis in these patients, the recommendations are based on studies which included a percentage of patients with cancer without primarily focusing on this high risk group.

Since patients with cancer present an increased risk of bleeding complications it is critical to evaluate the safety of thromboprophylaxis in the cancer group. Recent studies suggest a limited use of thromboprophylaxis in these patients.

The aim of this study is to evaluate the use, efficacy and safety of thromboprophylaxis in medical cancer patients hospitalized for an acute medical disease.

Design: observational, prospective study Primary end-point: incidence of major and clinically relevant non major bleeding during hospitalization Secondary endpoints: frequency of use, doses and contraindications for pharmacological thromboprophylaxis; venous thromboembolic events up to three months after discharge

ELIGIBILITY:
Inclusion Criteria:

* all patients with cancer hospitalized for an acute medical illness

Exclusion Criteria:

* current use of oral or parenteral anticoagulant treatment
* no informed consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer hospitalized for an acute medical illness
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2015-04; Primary Completion 2017-08 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Major bleeding and clinically relevant non major bleeding | Participants will be followed for the duration of hospital stay, an expected average of 1 week

SECONDARY OUTCOMES:
Venous thromboembolism | Participants will be followed up to 3 months after discharge, an expected average of 13 weeks
Minor bleeding | Participants will be followed for the duration of hospital stay, an expected average of 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Universita degli Studi G. d'Annunzio Chieti e Pescara, Chieti, Italy